CLINICAL TRIAL: NCT02008500
Title: COMPARISON OF CLINICAL EFFICACY OF A HERBAL AND A NON HERBAL MOUTHWASH ON DENTINAL HYPERSENSITIVITY: A TRIPLE MASKED RANDOMIZED CONTROLLED CLINICAL TRIAL
Brief Title: Comparison Of Clinical Efficacy Of A Herbal And A Non-Herbal Mouthwash On Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Collaborators: Himalaya Drug Company Research and Development, Makali, Bangalore, India (Unknown)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014
Record Dates: First submitted 2013-12-04; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Dentinal Hypersensitivity
Keywords: Dentinal Hypersensitivity; Gingival Recession; Visual Analogue Score
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Mouthwash Group (Placebo Comparator): Group 1 (placebo mouthwash group) contained 51 individuals
  Interventions: Other: placebo mouthwash
- Herbal Mouthwash Group (Active Comparator): Group 2 ( Herbal mouthwash) contained 52 individual
  Interventions: Other: Herbal Mouthwash
- Non Herbal Mouthwash Group (Sham Comparator): Group 3 (Non Herbal mouthwash) contained 50 individuals
  Interventions: Other: Non Herbal Mouthwash

INTERVENTIONS:
Other: placebo mouthwash — 15 ml placebo mouthwash prescribed and VAS score assessed at Baseline, 3 weeks, 6 weeks and 12 weeks
  Arms: Placebo Mouthwash Group
Other: Herbal Mouthwash — 15 ml Herbal mouthwash prescribed and VAS score assessed at Baseline, 3 weeks, 6 weeks and 12 weeks
  Arms: Herbal Mouthwash Group
Other: Non Herbal Mouthwash — 15 ml Non Herbal mouthwash prescribed and VAS score assessed at Baseline, 3 weeks, 6 weeks and 12 weeks
  Arms: Non Herbal Mouthwash Group

SUMMARY:
Aim of this study was to assess and compare the efficacy of a commercially available novel herbal mouthwash containing potassium nitrate on Dentinal Hypersensitivity (DH) compared to a placebo and non herbal potassium nitrate over a period of 12 weeks.

DETAILED DESCRIPTION:
A total of 120 subjects were divided into 3 groups randomly. Group 1 was given the placebo mouthwash, Group 2 was given the herbal mouthwash ( Hiora K, which contains potassium nitrate derived from Suryakshara plant) and Group 3 was given the non herbal mouthwash (Containing non herbal potassium nitrate). Sensitivity scores (VAS score) were recorded at baseline, 3 weeks, 6 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of DH caused by gingival recession or cervical erosion were selected at baseline. Subjects with a minimum 20 natural permanent teeth and at least two teeth with a VAS score of ≥4 were included in the study.

Exclusion Criteria:

* of teeth with caries, defective restorations, chipped teeth and deep periodontal pockets (probing depth >4 mm). Also, the subjects who had undergone periodontal surgery within the previous six months, and those with orthodontic appliances or bridge work that would interfere with evaluation were excluded. Subjects with the presence of occlusal overload or occlusal adjustment recently made in the tooth to be studied were also excluded. Subjects who had undertaken treatment with any product that could influence the DH of the patient in the 30 days prior to baseline were excluded. Also, the subjects with allergy to the ingredients used in the study or exhibiting any gross oral pathology, eating disorders, chronic disease, pregnancy and lactation, acute myocardial infarction within the past six months, uncontrolled metabolic disease, major psychiatric disorder, heavy smoking or alcohol abuse, any systemic disease or any disease requiring repeated or regular analgesia, anti-inflammatory drugs, or antihistamines were excluded from the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale score for Dentinal Hypersensitivity | Change in VAS score from Baseline to 12 weeks
  Based on a 10-cm VAS score which was used to measure tooth sensitivity, a pain-free response was allotted a score of zero whereas a score of 10 was given to subjects with excruciating pain or discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Avani R Pradeep, MDS, Principal Investigator — GDCRI, Bangalore, INDIA